CLINICAL TRIAL: NCT02303509
Title: A Randomised, Double-Blind, Placebo-Controlled, Single and Multiple Ascending Dose Study Evaluating The Safety/Tolerability, Pharmacokinetic and Pharmacodynamic Effects of UCB5857 in Healthy and Mild-to-Moderate Psoriatic Subjects
Brief Title: Study to Assess Safety, Tolerability, Pharmacokinetic & Pharmacodynamic Effect of UCB5857 in Healthy & Psoriatic Subject
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: UCB Pharma (Industry)
Collaborators: Parexel (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: PS0001; 2013-002323-42 (EudraCT Number)
Record Dates: First submitted 2014-11-25; First posted 2014-12-01 (Estimated); Last update posted 2014-12-01 (Estimated); Status verified 2014-11

CONDITIONS: Psoriasis
Keywords: Healthy Subjects; Mild to moderate Psoriasis; Subjects
MeSH Terms: conditions — Psoriasis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- UCB5857 Part 1 (Experimental): Part 1: Subjects assigned to UCB5857 or placebo single dose.
  Interventions: Drug: UCB5857 Part 1; Other: Placebo
- UCB5857 Part 2 (Experimental): Part 2: Subjects assigned to UCB5857 or placebo multiple doses.
  Interventions: Drug: UCB5857 Part 2; Other: Placebo

INTERVENTIONS:
Drug: UCB5857 Part 1 — Active substance: UCB5857
  Pharmaceutical form: Capsule
  Concentration: 1 mg, 5 mg, 10 mg or 15 mg
  Route of administration: Oral
  Arms: UCB5857 Part 1
Drug: UCB5857 Part 2 — Active substance: UCB5857
  Pharmaceutical form: Capsule
  Concentration: 5 mg, 8 mg, 15 mg
  Route of administration: Oral
  Arms: UCB5857 Part 2
Other: Placebo — Active substance: Placebo
  Pharmaceutical form: Capsule
  Concentration: Avicel PH 102, 50 mg
  Route of administration: Oral

SUMMARY:
To evaluate the safety and tolerability of UCB5857. Part 1 of the study explores single doses of the drug. Part 2 of the study explores giving the drug every day for 14 days. The study uses healthy and psoriasis subjects.

DETAILED DESCRIPTION:
This is a first-in-human (FIH), Phase 1, randomized, double-blind, placebo controlled, single center study designed to evaluate the safety/ tolerability, pharmacokinetics (PK), and pharmacodynamics (PD) of UCB5857 following oral administration of single ascending doses (SAD) in healthy subjects (Part 1) and multiple ascending doses (MAD) in healthy and mild-to-moderate psoriatic subjects (Part 2).

The primary objective of this study is to investigate the safety and tolerability of UCB5857 when given as single oral doses in healthy subjects and as ascending multiple oral doses in healthy subjects and mild-to-moderate psoriatic subjects.

ELIGIBILITY:
Inclusion Criteria:

* Subject is male or female, aged between 18 and 55 years (inclusive).
* Female subjects must have a negative serum pregnancy test at Screening, and be of nonchildbearing potential, defined as:

  * Being postmenopausal (for at least 2 years prior to Screening), verified by serum follicle-stimulating hormone (FSH) level >40 mIU/ mL at Screening, or
  * Having undergone complete hysterectomy, bilateral tubal ligation, and/ or bilateral oophorectomy, or
  * Being congenital sterile
* Male subject confirms that, during the study period and for a period of 3 months or 5 half lives after the last administration of the IMP (whichever is longer), when having sexual intercourse with a woman of childbearing potential, a method of highly effective contraception will be used (eg, condom + spermicide, and an additional contraceptive method used by the partner). Male contraception is not required if the male subject has undergone effective vasectomy >3 months prior to the study; however, his female partner must use a contraceptive method during the study period and for a period of 3 months or 5 half-lives after the last administration of the IMP (whichever is longer)
* Subject is of normal weight as determined by a body mass index (BMI) of between 18.0 and 30.0 kg/ m2 (inclusive), with a body weight of at least 50 kg (for healthy subjects only)
* Subject is in good physical and mental health, in the opinion of the Investigator, determined on the basis of medical history and general clinical examination at Screening
* Subject has clinical laboratory test results within the reference ranges of the testing laboratory. Subjects with isolated test results that are outside the specified ranges and that are deemed as clinically nonsignificant will be allowed at the discretion of the Investigator, following discussion with the Sponsor's Study Physician, excluding ALT, AST, alkaline phosphate and bilirubin, which have to be within normal range. If a subject has 1 isolated test result outside the specific range that is deemed clinically significant, rescreening may be allowed at the discretion of the Investigator, following discussion with the Sponsor's Study Physician
* Subject has BP and pulse rate within normal range in a supine position after 5 minutes rest (systolic BP: 90 to 140 mmHg, diastolic BP: 50 to 90 mmHg, pulse rate: 40 to 90 bpm). Results that are outside the specified ranges and that are deemed as clinically nonsignificant will be allowed at the discretion of the Investigator, following discussion with the Sponsor's Study Physician. If a subject has 1 isolated finding outside the specific range which is deemed clinically significant, rescreening may be allowed at the discretion of the Investigator, following discussion with the Sponsor's Study Physician
* Subject has a body temperature (oral or tympanic) between 35.0 and 37.5°C (95 and 99.5°F) inclusive
* Subject's ECG is considered "normal" or "abnormal" but clinically nonsignificant (as interpreted by the Investigator). If the subject has 1 isolated finding outside the specific range that is deemed potentially clinically significant, rescreening may be allowed at the discretion of the Investigator, following discussion with the Sponsor's Study Physician

In addition for the psoriatic subjects cohort

* Subject has a BMI at Screening <35 kg/ m2
* Subject has a confirmed diagnosis of mild-to-moderate plaque-type psoriasis for at least 6 months involving ≤10% of BSA (excluding the scalp)
* Subject has a minimum of 2 psoriatic lesions with at least 1 plaque in a site suitable for biopsies

Exclusion Criteria:

Subjects are not permitted to enroll in the study if any of the following criteria is met:

Healthy and psoriatic subjects

* Subject is an employee or direct relative of an employee of PAREXEL or the Sponsor
* Subject has participated in another study of an investigational medication (or a medical device) within the last 3 months or 5 half-lives of the study medication, whichever is longer, or is currently participating in another study of an investigational medication (or a medical device)
* Subject has made a blood donation (>400mL) or had a comparable blood loss (>350 mL) within the 3 months prior to first intake of study drug
* Subject tests positive for human immunodeficiency virus-1/2 antibody (HIV-1/2Ab), hepatitis B surface antigen, or hepatitis C virus antibody.
* Subject is not willing to avoid heavy physical exertion for 2 days before drug administration and during the study
* Subject has a history of alcohol and/or drug abuse up to 6 months before Screening
* Subject has an alcohol consumption of more than 21 units (males) or 14 units (females) of alcohol per week (1 unit of alcohol is equivalent to 10 mL ethanol; for example, 330 mL of 5 % alcohol by volume beer =1.7 units; 125 mL of 12 % wine =1.5 units: 50 mL of spirits with 40 % of alcohol by volume =2 units)
* Subject tests positive for alcohol and/or drugs (urine tests) at Screening or Day -1
* Subject has received any prescription (including hormonal replacement therapy) or nonprescription medicines, including over-the-counter (OTC) remedies, herbal, and dietary supplements (other than vitamins within recommended daily dose limits), within 21 days or 5 half-lives of the respective drug, whichever is longer, prior to Check-in (Day -1), other than occasional use of analgesics such as paracetamol (acetaminophen), ibuprofen, or intranasal corticosteroids for seasonal rhinitis
* Subject has consumed any grapefruit, grapefruit juice, or grapefruit-containing products, as well as St John's Wort-containing products, within 14 days prior to Check-in (Day -1)
* Subject has a known hypersensitivity to any components of the IMP
* Subject has current or past history of GI ulceration
* Subject is considered anti-immunoglobulin E (IgE) nonresponsive if CD63 induction on basophils is <10 %.
* Subject has cardiovascular or cerebrovascular disease, including hypertension, angina, ischemic heart disease, transient ischemic attacks, stroke, and peripheral arterial disease sufficient to cause symptoms and/ or require therapy to maintain stable status
* Subject has diabetes mellitus of any type requiring insulin
* Subject has unstable/poorly controlled Type 2 diabetes mellitus, defined as glycosylated hemoglobin type A1c (HbA1c) level ≥8.5 % or glucose intolerant
* Subject

  * Has an active infection (eg, sepsis, pneumonia, abscess)
  * Has history of latent, chronic, or recurrent infections (eg, tuberculosis, recurrent sinusitis, genital herpes, urinary tract infections) or at risk of infection (surgery, trauma, infection requiring antibiotics, history of skin abscesses) within 3 months prior to IMP administration
  * Has experienced a significant episode of gastroenteritis (defined as loose stools associated with abdominal pain and/ or fever) during the 7 days prior to IMP administration
  * When in doubt, the Investigator should confer with the Sponsor's Study Physician
* Subject has a history of positive tuberculosis (TB) test or evidence of possible TB or latent TB infection at Screening (interferon gamma release assay [IGRA] testing)
* Subject has received live attenuated vaccination within 3 months or any other type of vaccine within 4 weeks prior to Screening or intends to have such a vaccination during the course of the study
* Subject who has any of the following hematology values at Screening:

  * Hemoglobin; for women <11 g/ dL; for men <13 g/ dL
  * ANC <1.5x109/ L (<1500/ μL)
* Subject has an abnormality in the 12-lead ECG that, in the opinion of the Investigator, increases the risks associated with participating in the study. In addition any subject with any of the following findings will be excluded:

  * QTcF interval >450 ms in 2 of 3 ECGs.
  * Bundle branch blocks and other conduction abnormalities (other than mild first degree atrioventricular block) such that PR interval ≥220 ms
  * Irregular rhythms other than sinus arrhythmia or occasional, rare supraventricular or rare ventricular ectopic beats
  * In the judgment of the Investigator, T-wave configurations are not of sufficient quality for assessing QT interval duration
* Subject has active neoplastic disease or history of neoplastic disease within 5 years of Screening (except for basal or squamous cell carcinoma of the skin or carcinoma in situ that has been definitively treated with standard of care)
* Subject has any other acute or chronic illness which, in the opinion of the Investigator or the Sponsor's Study Physician, could pose a threat or harm to the subject
* Subject is legally institutionalized or has a mental health condition or related care provision (eg, guardianship) that would impede the subject from providing voluntary informed consent to participate in the study

Healthy subjects only

* The subject has used nicotine-containing products (including, but not limited to, cigarettes, pipes, cigars, chewing tobacco, nicotine patch, or nicotine gum) within 6 weeks prior to Check-in (Day -1) or anticipates an inability to abstain from these products for the duration of the study
* Subject has a high consumption of xanthine-containing products (≥300 mg of xanthine equivalent per day [1 cup of coffee ≈ 100 mg of caffeine; 1 cup of tea ≈ 30 mg of caffeine; 1 glass of cola ≈ 20 mg of caffeine]) Psoriatic subjects only
* Subject has received systemic nonbiologic psoriasis therapy (methotrexate [MTX], steroids, cyclophosphamide) or psoralen plus ultraviolet A (PUVA)/ultraviolet A (UVA) phototherapy within 4 weeks prior to Screening.
* Subject has received treatment with biologic agents within 12 months prior to the study

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 57 (Actual)
Dates: Start 2013-08; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events during the study | Day -1 to single dose Day 4 (Part 1) and Day -1 to multiple dose Day 18 (Part 2)

SECONDARY OUTCOMES:
Area under the plasma concentration-time curve from time 0 to the last quantifiable concentration (AUC(0-t)) | Pharmacokinetic samples will be taken predose and 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 24, 48 and 72 hours postdose on Day 1 (Part 1 and Part 2)
Area under the plasma concentration-time curve from time 0 to 24 hours (AUC(0-24)) | Pharmacokinetic samples will be taken predose and 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 24, 48 and 72 hours postdose on Day 1 (Part 1 and Part 2)
The area under the plasma concentration-time curve from time 0 to infinity (AUC) | Pharmacokinetic samples will be taken predose and 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 24, 48 and 72 hours postdose on Day 1 (Part 1 and Part 2)
The maximum observed plasma concentration of UCB5857 after single dosing, obtained directly from the observed plasma concentration-time curves (Cmax) | Pharmacokinetic samples will be taken predose and 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 24, 48 and 72 hours postdose on Day 1 (Part 1 and Part 2)
The time of occurrence of Cmax, obtained directly from the observed plasma concentration-time curves (tmax) | Pharmacokinetic samples will be taken predose and 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 24, 48 and 72 hours postdose on Day 1 (Part 1 and Part 2)
The apparent terminal half-life (t1/2) | Pharmacokinetic samples will be taken predose and 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 24, 48 and 72 hours postdose on Day 1 (Part 1 and Part 2)
The terminal elimination rate constant in plasma (λz) | Pharmacokinetic samples will be taken predose and 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 24, 48 and 72 hours postdose on Day 1 (Part 1 and Part 2)
The apparent volume of distribution after single dosing (Vz/F) | Pharmacokinetic samples will be taken predose and 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 24, 48 and 72 hours postdose on Day 1 (Part 1 and Part 2)
The apparent total body clearance after single dosing (CL/F) | Pharmacokinetic samples will be taken predose and 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 24, 48 and 72 hours postdose on Day 1 (Part 1 and Part 2)
Mean residence time (MRT) | Pharmacokinetic samples will be taken predose and 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 24, 48 and 72 hours postdose on Day 1 (Part 1 and Part 2)
Area under the plasma concentration-time curve from time 0 to the last quantifiable concentration (AUC(0-t)) | Pharmacokinetic samples will be taken predose and 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 24, 48 and 72 hours postdose on Day 14 (Part 2)
Area under the plasma concentration-time curve from time 0 to 24 hours (AUC(0-24)) | Pharmacokinetic samples will be taken predose and 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 24, 48 and 72 hours postdose on Day 14 (Part 2)
The time of occurrence of Cmax, obtained directly from the observed plasma concentration-time curves (tmax) | Pharmacokinetic samples will be taken predose and 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 24, 48 and 72 hours postdose on Day 14 (Part 2)
The apparent terminal half-life (t1/2) | Pharmacokinetic samples will be taken predose and 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 24, 48 and 72 hours postdose on Day 14 (Part 2)
The terminal elimination rate constant in plasma (λz) | Pharmacokinetic samples will be taken predose and 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 24, 48 and 72 hours postdose on Day 14 (Part 2)
Mean residence time (MRT) | Pharmacokinetic samples will be taken predose and 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 24, 48 and 72 hours postdose on Day 14 (Part 2)
The maximum observed plasma concentration of UCB5857 during steady state, obtained directly from the observed plasma concentration-time curves (Cmaxss) | Pharmacokinetic samples will be taken predose and 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 24, 48 and 72 hours postdose on Day 14 (Part 2)
The minimum observed plasma concentration of UCB5857 during steady state immediately before the next dose would be administered, obtained directly from the observed plasma concentration-time curves (Ctrough) | Pharmacokinetic samples will be taken predose and 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 24, 48 and 72 hours postdose on Day 14 (Part 2)
The apparent volume of distribution at steady state (Vzss/F) | Pharmacokinetic samples will be taken predose and 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 24, 48 and 72 hours postdose on Day 14 (Part 2)
The apparent total body clearance at steady state (CLss/F) | Pharmacokinetic samples will be taken predose and 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 24, 48 and 72 hours postdose on Day 14 (Part 2)
Accumulation factor based on AUC(0-24) (RAUC) | Pharmacokinetic samples will be taken predose and 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 24, 48 and 72 hours postdose on Day 14 (Part 2)
Accumulation factor based on Cmax (R(Cmax)) | Pharmacokinetic samples will be taken predose and 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 24, 48 and 72 hours postdose on Day 14 (Part 2)
Time independency factor (TI) | Pharmacokinetic samples will be taken predose and 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 24, 48 and 72 hours postdose on Day 14 (Part 2)
Total amount of drug excreted in urine from time 0 to time t (Ae(0-t)) | Urine pharmacokinetic samples will be taken predose and 0 - 5 hours, 5 - 10 hours, 10 - 24 hours, 24 - 48 hours, 48 - 72 hours postdose on Day 1 (Part 1 and Part 2) and on Day 14 (Part 2)
Renal clearance (CLr) | Urine pharmacokinetic samples will be taken predose and 0 - 5 hours, 5 - 10 hours, 10 - 24 hours, 24 - 48 hours, 48 - 72 hours postdose on Day 1 (Part 1 and Part 2) and on Day 14 (Part 2)
Fraction of drug excreted in urine (Fe) | Urine pharmacokinetic samples will be taken predose and 0 - 5 hours, 5 - 10 hours, 10 - 24 hours, 24 - 48 hours, 48 - 72 hours postdose on Day 1 (Part 1 and Part 2) and on Day 14 (Part 2)
Basophil degranulation | Samples will be taken predose, 0.5, 1, 2, 4, 6, 8, 10, 24 hours postdose on Day 1 (Part 1 and Part 2) and predose, 0.5, 1, 2, 4, 6, 8, 10, 24, 48 hours postdose on Day 14 (Part 2)

CONTACTS AND LOCATIONS:
Overall Officials: UCB, Cares, Study Director — 1-877-822-9493
Locations (1):
- 001, Harrow, United Kingdom